CLINICAL TRIAL: NCT00328757
Title: Regular Versus Liquid Diet as the First Meal in Patients Undergoing Major Abdominal Gynecologic Cancer Operation: A Randomized Controlled Trial
Brief Title: Safety of Regular Diet as the First Meal in Patients Who Underwent Surgical Treatment for Gynecologic Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Before starting the recruitment process, new data from literature were available. The investigators considered that this study was no longer needed.
Sponsor: Chiang Mai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OF-01
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Gynecologic Neoplasms
Keywords: gynecologic cancer; cervical cancer; ovarian cancer; endometrial cancer; radical abdominal hysterectomy; pelvic lymphadenectomy; surgical staging; postoperative feeding; Early-stage gynecologic cancer patients
MeSH Terms: conditions — Genital Neoplasms, Female; Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms | interventions — Diet

INTERVENTIONS:
Behavioral: Regular diet as the first postoperative meal

SUMMARY:
The purpose of this study is to determine whether it is safe to give a regular diet as the first postoperative meal in patients who underwent surgical treatment for clinically early-stage gynecologic cancer.

DETAILED DESCRIPTION:
Paralytic ileus, a temporary inhibition of bowel motility, is believed to follow all abdominal surgery. Surgeons have customarily withheld postoperative oral intake until the return of bowel function as evidenced by a presence of bowel sound, a passing of flatus/stool, and a feeling of being hungry. The major concern has been that early oral intake would result in vomiting from severe paralytic ileus with subsequent aspiration pneumonia, wound dehiscence, and anastomotic leakage. Recently, the practice of delayed postoperative oral intake has been challenged by evidence from extensive gastrointestinal physiologic studies that examine contractile activity of the intestine. These data have suggested that the concept of postoperative ileus as paralysis of the entire bowel with complete absence of any functional contractile activity is misleading. If postoperative ileus takes place, it is usually transient and not significant clinically. Several possible clinical benefits of early feeding after surgery exist that include better wound healing, postoperative stress ulcer prevention, reduced sepsis, improved sense of well being, shorter length of hospital stay, and cost saving. Currently, the practice of early administration of liquid diet after surgery has become widely accepted. For early regular diet administration, the proposed additional benefits would be lesser risk of aspiration, faster recovery of intestinal motility, and better nutritional status. Patients who had surgery as a treatment for gynecologic cancer deserve special attention in this regard as they generally have higher risk of developing postoperative ileus due to extensive and/or multiple intraabdominal surgical procedures including radical hysterectomy, pelvic lymph node dissection, and surgical staging procedures. At the same time, this is the group of patients that would benefit most from the aforementioned positive effects of early regular diet feeding.

Comparisons: Regular versus liquid diet as the first postoperative meal on the first day after surgery for clinically early-stage gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinically early-stage gynecologic cancer patients who underwent standard abdominal surgery as a primary treatment of their diseases

Exclusion Criteria:

* Peritonitis
* Perioperative hyperalimentation
* Bowel surgery (except appendectomy)
* Bowel obstruction
* History of bowel surgery or inflammatory bowel syndromes
* History of abdominal/pelvic radiotherapy
* Need for continued postoperative endotracheal tube or naso/orogastric tube placement
* Need for postoperative Intensive Care Unit (ICU) administration
* Pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2006-05; Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically significant postoperative ileus

SECONDARY OUTCOMES:
Patient's satisfaction
Other postoperative complications
Time to first flatus
Amount of meal taken
Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, M.D., Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Muang Chiangmai, Chiang Mai, Thailand

REFERENCES:
- [Background] Jeffery KM, Harkins B, Cresci GA, Martindale RG. The clear liquid diet is no longer a necessity in the routine postoperative management of surgical patients. Am Surg. 1996 Mar;62(3):167-70. PMID 8607572
- [Background] Patolia DS, Hilliard RL, Toy EC, Baker B. Early feeding after cesarean: randomized trial. Obstet Gynecol. 2001 Jul;98(1):113-6. doi: 10.1016/s0029-7844(01)01387-4. PMID 11430967
- [Background] MacMillan SL, Kammerer-Doak D, Rogers RG, Parker KM. Early feeding and the incidence of gastrointestinal symptoms after major gynecologic surgery. Obstet Gynecol. 2000 Oct;96(4):604-8. doi: 10.1016/s0029-7844(00)00957-1. PMID 11004367